CLINICAL TRIAL: NCT03561935
Title: Outcome of Medical Treatment for Idiopathic Premature Ventricular Complexes - Beta-blocker vs Ic Antiarrhythmic Agent; Randomized Controlled Trial
Brief Title: Beta-blocker vs. Ic Antiarrhythmic Drug for PVC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Yong Seog Oh (Other)
Responsible Party: Sponsor-Investigator, Yong Seog Oh, professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PVC study
Record Dates: First submitted 2017-04-24; First posted 2018-06-19 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Premature Ventricular Complex
MeSH Terms: conditions — Ventricular Premature Complexes | interventions — Propafenone; 1-indenol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propafenone group (Experimental): Prescribtion of propafenone for the management of premature ventricular complex
  Interventions: Drug: Propafenone
- Indenol group (Active Comparator): Prescribtion of indenol for the management of premature ventricular complex
  Interventions: Drug: Indenol

INTERVENTIONS:
Drug: Propafenone — prescribing propafenone for the management of premature ventricular complex
  Arms: Propafenone group
Drug: Indenol — prescribing indenol for the management of premature ventricular complex
  Arms: Indenol group

SUMMARY:
The standard medical therapy of idiopathic premature ventricular complex consists of beta blocker and Ic antiarrhythmic agent. However, the difference in the efficacy of two drugs has not been well investigated. This prospective randomized study aimed to compare the efficacy of beta-blocker and Ic antiarrhythmic agent in the treatment of symptomatic patients with idiopathic premature ventricular complex.

DETAILED DESCRIPTION:
A premature ventricular complex is frequently observed in routine clinical practice and patients without structural heart disease occasionally have benign outcomes. The initial therapy of symptomatic premature ventricular complex is medical treatment with beta-blocker, calcium channel blocker or antiarrhythmic agents. However, no large prospective study has been performed to identify the difference in the efficacy between drugs. The current study was designed to compare the efficacy between beta-blocker and class Ic antiarrhythmic agent. Patient with symptomatic PVC more than 6000 episode per 24 hours is included. Exclusion criteria are evidence of structural heart disease, coronary heart disease, significant bradycardia or use of a concomitant antiarrhythmic agent. Patients are randomized into beta-blocker group (propranolol) and Ic antiarrhythmic agent group (propafenone). Response to the drug is evaluated after 2 months from randomization by 24 hours Holter and questionnaire. The primary endpoint is more than 80% PVC reduction or PVC burden less than 300 beats per 24 hours. The secondary endpoint is patient's symptom evaluated by questionnaire and the number of PVCs measured in 24 hours Holter.

ELIGIBILITY:
Inclusion Criteria:

* over 19 years old >6000 PVCs/24hrs

Exclusion Criteria:

* Left ventricular ejection fraction <50% or Significant valvular disease (≥moderate) History of coronary artery disease Use of a concomitant antiarrhythmic agent Significant bradycardia

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2019-06-01 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in PVC frequency on 24hrs holter | two months after randomization
  PVC reduction of >80% or <300 beats/day

CONTACTS AND LOCATIONS:
Overall Officials: Yong-Seog Oh, MD,PhD, Principal Investigator — The Catholic University of Korea
Locations (1):
- Seoul St Mary's Hospital, Seoul, Seo Ch-gu, South Korea